CLINICAL TRIAL: NCT05023993
Title: The Effect of Exercise and Nicotinamide Riboside on Muscle Health and Insulin Resistance in Adult Survivors of Childhood Cancer With Prediabetes: A Pilot Feasibility Study
Brief Title: The Effect of Exercise and Nicotinamide Riboside Muscle Health and Insulin Resistance in Survivors of Childhood Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20676; NCI-2021-02807 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20676 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2021-08-04; First posted 2021-08-27 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm; Prediabetes
MeSH Terms: conditions — Hematologic Neoplasms; Prediabetic State | interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (home exercise) (Active Comparator): Patients complete 18 home exercise sessions over 30 minutes each, 3 days per weeks for 6 weeks.
  Interventions: Other: Exercise Intervention
- Arm II (home exercise, nicotinamide riboside) (Experimental): Patients complete home exercise as in Arm I. Patients also receive nicotinamide riboside PO daily for 6 weeks.
  Interventions: Other: Exercise Intervention; Dietary Supplement: Nicotinamide Riboside

INTERVENTIONS:
Other: Exercise Intervention — Complete home exercise
Dietary Supplement: Nicotinamide Riboside — Given PO
  Other Names: Niagen; NR
  Arms: Arm II (home exercise, nicotinamide riboside)

SUMMARY:
This trial studies the effect of exercise and nicotinamide riboside on muscle health and insulin resistance in adult survivors of childhood cancer with prediabetes (elevated blood sugar level that is not high enough to be considered diabetes). Nicotinamide riboside is a dietary supplement which is similar to vitamin B3. Information collected in this study may help the future development of regimens to improve metabolic outcomes such as muscle health and insulin resistance (when the body is not normally responding to insulin) in childhood cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate the feasibility of conducting a home exercise and nutrition intervention in childhood cancer survivors (CCS) with a history of prediabetes.

EXPLORATORY OBJECTIVES:

I. Describe the association between patient demographics and treatment exposures and subsequent hyperglycemia and skeletal muscle health in childhood cancer survivors.

II. Describe the effect of exercise with or without nicotinamide riboside (NR) on hyperglycemia and skeletal muscle health in CCS with a history of prediabetes.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients complete 18 home exercise sessions over 30 minutes each, 3 days per weeks for 6 weeks.

ARM II: Patients complete home exercise as in Arm I. Patients also receive nicotinamide riboside orally (PO) daily for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* History of childhood cancer
* History of prediabetes (HbA1c 5.7-6.4%)
* In remission at time of enrollment
* Time between completion of cancer-directed therapy and study entry: >= 6 months
* At least 18 years of age at time of enrollment
* Able to access online exercise program at home
* Ability to tolerate the prescribed resistance exercise program
* English-speaking
* Able to understand and sign the study specific informed consent form (ICF)

Exclusion Criteria:

* Taking a nicotinamide adenine dinucleotide (NAD)+ precursor in the two weeks prior to enrollment
* Currently taking medication for hyperglycemia or diabetes
* Females who are pregnant or planning to become pregnant
* Currently recovering from an injury
* Contraindication to magnetic resonance imaging (MRI)
* Pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-06-23 (Actual); Primary Completion 2026-09-21 (Estimated); Study Completion 2026-09-21 (Estimated)

PRIMARY OUTCOMES:
Feasibility of a nutrition and exercise program in childhood cancer survivors (CCS) | Up to 6 weeks
  The current protocol will be considered feasible if:
  1. >= 50% of eligible patients that are approached for participation enroll onto the study,
  2. >= 70% of enrolled participants successfully complete all study assessments (i.e. physical function tests, blood draw, imaging, and questionnaires at baseline and 6 weeks, and
  3. Enrolled participants demonstrate >= 70% compliance with prescribed exercise and nicotinamide riboside.
  Feasibility measures 2 and 3 will be assessed for the entire group of 20 subjects as a whole.

CONTACTS AND LOCATIONS:
Overall Officials: Rusha Bhandari, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States